CLINICAL TRIAL: NCT05549414
Title: Pivotal Study of Proton Radiotherapy Treatments Using Fixed Beam Chair-Based Delivery System
Acronym: PPTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: P-Cure (Industry)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PC001
Record Dates: First submitted 2022-08-31; First posted 2022-09-22 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-03

CONDITIONS: Thoracic Cancer; Pancreatic Cancer Non-resectable; Brain Cancer; Head Cancer; Neck Cancer
MeSH Terms: conditions — Brain Neoplasms; Head and Neck Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients with locally recurrent, previously irradiated thoracic cancer (Experimental): Prospective study shall evaluate treatment efficacy, toxicity, QOL and plan parity in patients with recurrent thoracic cancer previously irradiated, undergoing proton radiation therapy
  Interventions: Device: Proton Radiation
- Patients with recurrent Head and Neck, Brain and Spinal Cord tumors, indicated for re- irradiation (Experimental): The prospective study shall evaluate treatment Efficacy, Toxicity, Quality of Life (QOL), and plan parity in adult patients with recurrent Head and Neck and Brain cancer undergoing proton radiation therapy
  Interventions: Device: Proton Radiation
- Patients with unresectable pancreatic cancer (Experimental): This prospective study shall evaluate treatment feasibility utilizing the CBGS for unresectable pancreatic cancer with concurrent chemotherapy
  Interventions: Device: Proton Radiation

INTERVENTIONS:
Device: Proton Radiation — Proton beam radiotherapy, first proposed by Robert Wilson at Harvard University in 1946, utilizes an energetic beam of ionized hydrogen nuclei (protons) directed at the tumor volume to effect DNA damage of the targeted cells. Today, there are hundreds of proton treatment centers worldwide and it is considered standard treatment for certain malignancies and/or clinical scenarios
  Other Names: p-cure PROTON RADIATION SYSTEM; Proton Beam Radiation Therapy; Quality-of-Life Assessment

SUMMARY:
This study with Chair-Based, Gantry-less Proton System (CBGS) (aka P-CURE Proton Beam Therapy System or Fixed Beam Chair-based Delivery System) is composed of 3 arms, as following:

ARM1: Patients with locally recurrent, previously irradiated thoracic cancer indicated for re- irradiation.

ARM2: Patients with recurrent Head and Neck, Brain and Spinal Cord tumors, indicated for re- irradiation.

ARM3: Patients with unresectable pancreatic cancer.

The primary objectives of the study for all arms are: 1. to describe the efficacy (local control after 3 month) and acute toxicity for patients treated with a fully-integrated CBGS and (2) to compare treatment plans between the fully-integrated CBGS and Photon therapy defined for each patient, based upon OAR sparing for comparable target coverage.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven malignancy
* Treatment planning analysis shows advantage to proton over photon treatments
* both malignancies (such as thoracic tumors) as well as metastatic lesions (such as metastatic breast cancer or colorectal cancer to the lungs) are allowed
* Patient must have CT confirmation of the tumor
* Patients must have a life expectancy of > 6 months
* Patients must have measurable disease to be treated with proton radiation (minimum tumor dimension at least 10 mm on CT imaging).
* Patients must be a candidate for definitive radiation dose
* There are no limits on prior therapy. Patients are allowed to have prior chemotherapy and surgery. Patients are allowed to have concurrent chemotherapy with radiation treatment. Patients are allowed to have chemotherapy or surgery after radiation treatment

Exclusion Criteria:

1. Severe, active co-morbidity, defined as follows:

   1. Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
   2. Transmural myocardial infarction within the last 6 months
   3. Chronic obstructive pulmonary disease exacerbation or other respiratory illness other than the diagnosed lung cancer requiring hospitalization or precluding study therapy within 30 days before registration
   4. Acquired immune deficiency syndrome (AIDS) based upon current CDC definition (protocol may be significantly immunosuppressive endangering AIDS patients)
2. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
3. Patients with life expectancy < 6 months
4. Patients that participate in another, active clinical trial carried out concurrently with this protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Local Control | 3 months
  The duration of local control will be measured from the start date of protocol radiation until the date of progressive disease. Local control will be determined based on RECIST Criteria Version 1.1.
Acute Toxicity | 3 months
  Incidence of treatment-related grade 3-5 adverse events, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
Treatment Plan Comparison between Chair Based Proton System and Photon therapy | 3 months
  Analysis and comparison of dose volume histograms (DVHs) and isodoses for each modality

SECONDARY OUTCOMES:
Progression Free Survival | 2 years
  The time from study registration until the first occurrence of local, regional, or distant progression, or death from any cause, or until last follow-up
Overall Survival | 2 years
  The time from study registration until death or last follow-up
Long-term Toxicity | 2 Years
  Incidence of treatment-related grade 3-5 adverse events, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
Quality of Life | 2 years
  Lung Cancer Patients: FACT-Lung and EQ-5D Head and Neck Patients: EORTC QLQ-C30 and the EORTC QLQ-H&N35 Pancreas Patients: Quality of Life assessment using Patient Reported Outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Ein Karem, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No